CLINICAL TRIAL: NCT01722578
Title: Efficacy of Intravenous 'L-ornithine L-aspartate' in Reversal of Overt Acute Hepatic Encephalopathy in Patients With Liver Cirrhosis: a Prospective, Randomized, Double-blind, Placebo Controlled Trial
Brief Title: L-ornithine L-aspartate in Overt Hepatic Encephalopathy
Acronym: HEAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dayanand Medical College and Hospital (Other)
Responsible Party: Principal Investigator, Prof. Sandeep S Sidhu, Professor, Dayanand Medical College and Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEAL-123
Record Dates: First submitted 2012-10-30; First posted 2012-11-07 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Cirrhosis of Liver; Hepatic Encephalopathy
Keywords: Cirrhosis; Encephalopathy; L-ornithine L-aspartate
MeSH Terms: conditions — Fibrosis; Hepatic Encephalopathy; Brain Diseases | interventions — ornithylaspartate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-ornithine L-aspartate (Experimental): L-ornithine L-aspartate (6 ampules, each ampule containing 5 grams of the drug in 10 ml solution) to be diluted in 440 ml of Dextrose 5% (to make a total of 500 ml of solution), as intravenous infusion at the rate of 21 ml/hour, over 24 hours, for 5 days
  Interventions: Drug: L-ornithine L-aspartate
- Placebo (sterile water) (Placebo Comparator): Placebo (sterile water, 6 ampuoles of 10 ml each) diluted in 440 ml of Dextrose 5%, as intravenous infusion at the rate of 21 ml/hour, over 24 hours, for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-ornithine L-aspartate — L-ornithine L-aspartate (6 ampules, each ampule containing 5 grams of the drug in 10 ml solution) to be diluted in 440 ml of Dextrose 5% (to make a total of 500 ml of solution), as intravenous infusion at the rate of 21 ml/hour, over 24 hours, for 5 days
  Other Names: Hepamerz
  Arms: L-ornithine L-aspartate
Drug: Placebo — Placebo (sterile water, 60 ml) diluted in 440 ml of Dextrose 5%, as intravenous infusion at the rate of 21 ml/hour, over 24 hours, for 5 days
  Arms: Placebo (sterile water)

SUMMARY:
Hepatic encephalopathy (HE) is a potentially reversible functional disorder of the brain with neurological and psychiatric symptoms. HE occurs in up to 70% of patients with cirrhosis at some time during the course of disease. The chief neurotoxin implicated in the development of HE is ammonia. An important aim of treatment of HE is the reduction of the ammonia in the body by lowering the amount of ammonia produced and increasing its detoxification. Enteric production of ammonia can be decreased by non-absorbable disaccharides such as lactulose and antibiotics such as rifaximin. L-ornithine- L-aspartate (LOLA), the salt of the natural amino acids ornithine and aspartate acts through the mechanism of substrate activation to detoxify ammonia. In clinical trials, LOLA has shown a statistically significant effect with respect to reduction in HE grade, reduction of blood ammonia concentration and positive effects on psychomotor function in patients of cirrhosis with minimal HE and overt chronic Grade I HE, as compared to placebo. However, there is lack of data on the efficacy of LOLA in patients with overt acute hepatic encephalopathy which is one of the major causes of hospital admissions and resource utilization in decompensated cirrhotics. Each admission for HE causes a major financial loss to the family and financial burden on the society. Any drug which decreases the hospital stay by rapidly improving HE, will clearly lead to decreased hospital costs to the individual and the society as a whole. Hence, such a trial is a national priority. The investigators hypothesize that LOLA, if added to the standard treatment of overt acute HE (i.e lactulose), may lead to a faster recovery and decrease in hospital stay of these patients. In this prospective, randomized, placebo controlled trial, the investigators aim to evaluate the efficacy of intravenous L-ornithine, L-aspartate in reversal of overt acute hepatic encephalopathy in patients with liver cirrhosis.

DETAILED DESCRIPTION:
A. Introduction and Review of literature

Hepatic encephalopathy (HE) is broadly defined as an alteration in mental status and cognitive function occurring in presence of liver failure. The clinical picture of HE arises as a complication of chronic and, more rarely, acute liver disease. HE occurs in up to 70% of patients with cirrhosis at some time during the course of their disease (1,2). It is characterized by personality changes, intellectual impairment and a depressed level of consciousness. HE may be clinical unapparent (minimal HE) detected by abnormal neuropsychometric or neurophysiological tests (3). The common presentation is overt HE which occurs in patients with advanced cirrhosis with portal-systemic collateral circulation. Episodes of HE in patients with cirrhosis are induced by precipitating factors, like dehydration, hypokalemia, large protein intake, gastrointestinal bleeding, constipation, infections, use of psychotropic drugs, alcohol intake or acute liver injury (hepatitis).

Pathogenesis of hepatic encephalopathy In patients with liver cirrhosis, increasing structural replacement of hepatocytes with connective tissue leads to the loss of functioning hepatic parenchymal tissue and a reduction in the detoxification capacity of the liver. In addition, developing portal hypertension leads to the formation of a collateral circulation through which non-detoxified blood can by-pass the liver to reach the systemic circulation. Both these mechanisms contribute to the neurotoxins present in portal vein blood reaching the brain via the systemic circulation. A number of neurotoxins have been implicated in the pathogenesis of HE with ammonia being the most important (4,5). Fundamental conceptual advances in our understanding of hepatic encephalopathy have confirmed the central role of ammonia in the pathogenesis of portosystemic encephalopathy. Ammonia disrupts the function of neurones and astrocytes, giving rise to the symptoms of hepatic encephalopathy.

Classification/Grading of HE can be classified as type A (in Acute Liver Failure), B (in Portosystemic shunts without intrinsic liver disease) and C (patients of cirrhosis with portal hypertension/or portosystemic shunts) (5,6). In cirrhotics, the type C HE is further classified into Episodic, Persistent and Minimal HE. Chronic persistent overt HE patients are those who can be relatively stable with little day to day fluctuation in their mental status. Episodic (Unstable) HE patients are defined as those who were previously stable, but who over hours and possibly days develop clinically discernible features of HE, requiring medical attention and hospitalization. Minimal HE is clinically inapparent and detected by abnormal neuropsychometric or neurophysiological tests (3).

A precise gradation of HE is essential to prognosticate and plan an appropriate approach to treatment. According to the severity, HE has been traditionally divided into four stages based on alterations in the state of consciousness, intellectual function, behaviour, and neuromuscular signs (West Haven scale) (5).

A new classification has been recently proposed called the SONIC classification (7). This was necessary because the differentiation between minimal and Grade I HE is not reliable, but there is good inter-rater reproducibility in the identification of Grade II HE. It was suggested that patients with minimal HE and Grade I HE should be grouped together. It stresses that worsening cognitive function is continuum rather than categorical as emphasized in the Vienna 11th World Congress. It classifies patients with cirrhosis as being unimpaired and impaired neurocognitive function. Impaired cognitive function is subdivided into Covert HE (Minimal HE and Grade I HE) and Overt HE (Grades II-IV). It is thus inclusive of the West Haven criteria, yet emphasizes continuity as opposed to being categorical. The neurocognitive function of impaired, unstable patients can fluctuate from acute confusional syndrome to coma (Grades I to IV). They are the so called Type C- episodic HE patients.

Therapy of hepatic encephalopathy The main objective of therapy of HE is to (a) decrease intestinally derived toxins produced by excessive bacterial activity and decrease ammonia production or (b) increase ammonia detoxification (1,2,8,9).

1. Decrease ammonia production:

   Enteric production of ammonia can be decreased by non-absorbable disaccharides such as lactulose or lactitol and non-absorbable antibiotics such as rifaximin. Lactulose/lactitol pass through the small bowel undigested. In the colon, bacteria degrade lactulose to various organic acids (e.g. lactic acid, acetic acid) with subsequent lowering of colonic pH. The mode of ammonia lowering may involve bacteriostatic effects, cathartic effects, or enhancement of conversion of ammonia to ammonium with excess hydrogen ion. Presumably ammonium is then excreted into the feces and eliminated (9, 10). Lactulose remains the main stay of therapy of overt HE, despite the paucity and inconsistency of clinical trials demonstrating its efficacy (11). The dosage should be adjusted to accomplish two to three soft bowel movements each day. Lactulose can be given through a nasogastric tube or through retention enemas. The usual dose is 30-120 ml each day in divided doses. Stool pH should be below six. Side effects include bloating and flatulence. Severe diarrhea with dehydration and hyperglycemia and acidosis occurs if the dosage is too high.

   Non absorbable antibiotics neomycin, metronidazole, and paromomycin are traditional antibiotics for the treatment of HE (12). Due to ototoxic and nephrotoxic side effects, neomycin is now used infrequently. Metronidazole does not cause much side effects but therapy should not extend beyond two weeks to avoid neuropathy. More recently rifaximin has demonstrated to be as good as lactulose (13) or lactitol (14, 15) for patients with hepatic encephalopathy.
2. Increase ammonia detoxification:

Levels of ammonia can be decreased by detoxification. L-ornithine- L-aspartate (LOLA), the salt of the natural amino acids ornithine and aspartate acts through the mechanism of substrate activation to detoxify ammonia. Detailed mechanism of action and clinical trials on LOLA are discussed below.

L-ornithine- L-aspartate (LOLA):

L-ornithine- L-aspartate (LOLA) is the salt of the natural amino acids ornithine and aspartate.

1. Mechanism of action:

   LOLA stimulates the urea cycle (which metabolizes ammonia to urea) in the liver (16,17). In the periportal hepatocytes that synthesize urea, ornithine serves as an activator of ornithine transcarbamoylase and carbamoyl phosphate synthetase. In addition, ornithine can acts as a substrate for urea genesis. Hence, LOLA can activate the periportal urea cycle in the liver. Aspartate and ornithine, after conversion to alpha- ketoglutarate, also serves as carbon sources for perivenous glutamine synthesis. In the skeletal muscle, LOLA upregulates glutamine synthesis by substrate provision for glutamine synthetase, although decreased muscle mass in cirrhosis does not allow this synthesis to be significant. Ammonia is consumed during urea formation and glutamine synthesis, and thereby LOLA decreases blood ammonia levels. Urea and glutamine (after further metabolism) can be excreted via the kidneys. LOLA thus activates the two important metabolic pathways in the human body for the detoxification of ammonia. In cirrhosis, there is some remaining liver cell mass that retains capacity to detoxify ammonia as opposed to acute liver failure.
2. Trials of LOLA in Hepatic encephalopathy:

   LOLA has been used for many years for the treatment of HE in cirrhosis of the liver, especially minimal and overt chronic low grade HE. The clinical efficacy of LOLA has already been comprehensively investigated and reported in therapeutic observations, clinical trials (16, 18-25) and meta-analysis (26,27). In these studies, the use of LOLA as infusion, oral administration or a combination of the two, was documented in patients with mild to severe liver insufficiency. LOLA showed a statistically significant effect with respect to an improvement in mental state (reduction in the HE grade), increased detoxification (reduction of the ammonia concentration in the blood) and positive effects on psychomotor function (reduction of time required in the number connection test) in Minimal Hepatic Encephalopathy and overt chronic Grade I-II Hepatic Encephalopathy, and acute overt HE. With these findings, evidence-based medicine criteria for demonstrating efficacy have been fulfilled.

   In a recent randomized placebo controlled study conducted at Karachi (25), patients with acute HE were randomized to receive LOLA or placebo. NCT-A, ammonia level, clinical grade of HE and duration of hospitalization were assessed. Improvement in HE was higher (n=40, 66.7%) in LOLA group (n=28, 46.7%, p=0.027). Duration of hospitalization was lower in LOLA group compared to placebo (p=0.025). No side effects were observed in either group.
3. Adverse effects of LOLA L-ornithine- L-aspartate is usually well tolerated (18-25). No serious adverse events have been reported so far in clinical trials. The various adverse events reported in about 14% patients treated with LOLA include:

   1. Nausea
   2. Vomiting
   3. Fatigue

B. Materials and Methods

1. Study design and setting:

   This will be a prospective, randomized, double blind, placebo controlled interventional study.

   The study will be conducted on patients of cirrhosis admitted with overt HE in the Department of Gastroenterology, Dayanand Medical College and Hospital, Ludhiana and Department of Hepatology, GB Pant Hospital, New Delhi. Informed consent shall be taken from the nearest relative of the patient for enrollment in the trial.

   The study shall be presented for approval to the Institutional Ethics Committee prior to the enrollment of patients into the study. It shall be registered with Clinical Trial Registry, India and the ClinicalTrials.gov registry.
2. Study population:

   Inclusion and exclusion criteria have been mentioned elsewhere.
3. Study Methods:

   Assignment: Consecutive patients diagnosed to have acute overt HE will be randomized into two groups (group A and B) using sealed opaque envelopes containing computer-generated random numbers. There shall be no restriction, blocking or stratification of the randomization sequence. The research coordinator who will generate the sequence shall have no role in recruitment, treatment, or assessment of patients.

   Masking: Sequentially numbered boxes containing identical LOLA or placebo ampoules, according to the allocation sequence will ensure allocation concealment. The numbering of the boxes will be done by research coordinator, and concealed from the treating consultants. All study personnel will be blinded to the treatment assignment (placebo or LOLA) for the duration of the study. Placebo and LOLA will be similar in appearance and in the mode of administration. The code of the allocation sequence will remain with the research coordinator. It will be revealed only after the recruitment, data collection and analysis of results has been carried out. The coordinator will not have any access to the patients involved in the study.

   Randomization implementation: Enrollment of patients, assessing eligibility and obtaining informed consent will be carried out by one of the investigators (S.S. Sidhu or O. Goyal, BC Sharma) Study Intervention: The patients will be randomized to receive either placebo or LOLA at dose of 30 grams daily, by intravenous infusion over 24 hours. (The study drugs and placebo will be provided by Win Medicare Pvt Ltd., 1400, Modi tower, 98, Nehru Place, New Delhi- 110019). LOLA will be supplied as ampoules (each ampoule containing 5 grams LOLA in 10 ml clear solution). Six ampoules (i.e 30 g of LOLA) will be infused over 24 hours. The placebo vials (10 ml sterile water in each vial) will be identically supplied and infused. The dose of LOLA (30 g in 24 hours) was based on previous studies, showing the efficacy of this dose in decreasing ammonia levels (17,26,28). Both groups shall receive treatment for 5 days. Patients in both the groups who continue to have hepatic encephalopathy at the end of study period (5 days), will receive standard of care treatment, and would be counseled about liver transplant.
4. Laboratory tests:

   Biochemical tests: Hemogram, blood glucose, liver function tests, prothrombin time, serum electrolytes, blood urea and serum creatinine will be done at baseline, and at 2nd and 5th day of treatment, or earlier if indicated. Serum AFP will be done at admission. Serum cytokine levels (Interleukin 1, 6, 10 and TNF-alpha) levels will be done at baseline and after 5 days of treatment.

   Microbiologic tests: A diagnostic paracentesis will be done in all patients with ascites, at baseline, to diagnose Spontaneous Bacterial Peritonitis. A repeat cell count (Total and differential) shall be done on day 5 with patients diagnosed to have Spontaneous Bacterial Peritonitis. Blood culture, urine culture, cultures of aspirates from endotracheal tubes in ventilated patients for aerobic and anerobic bacteria, and fungi shall be done. A chest radiograph shall also be done.

   Ammonia estimation: Fasting venous ammonia levels will be estimated by using the blood ammonia meter (PocketChem BA) at baseline and then daily for the next 5 days. The PocketChem BA ammonia meter is an apparatus for quick bedside blood ammonia estimation. It has been shown to have acceptable precision, adequate linearity, and satisfactory agreement with a enzymatic reference method commonly used in clinical laboratories (29).

   Measurement Principle: The PocketChem BA measures blood ammonia based on the micro-diffusion method. When the blood sample (20 microlitre) is applied to the sample-receiving layer of the test area on the test strip, the alkaline buffer agent (borate buffer) impregnated in the layer dissolves making the specimen alkaline. The ammonium ions in the specimen are gasified by the alkaline state into ammonia gas. The ammonia gas passes through the pores of the spacer to the indicator (bromocresol green) triggering color development. As the degree of color development is proportional to the concentration of ammonia gas produced, the blood ammonia level is quantitatively determined by measuring the color.

   Tests for etiologic evaluation: Etiology of cirrhosis will be taken as alcohol if there is a history of significant alcohol intake (40-60gm/day for females, and 60-80 gm/day for males for 10 years). Each patient will be tested for Hepatitis B surface antigen (HbsAg) and Anti-hepatitis C (HCV) antibody using a third generation commercial ELISA. Wherever indicated, autoimmune hepatitis will be diagnosed using antinuclear antibody, anti-smooth muscle antibody and anti-LKM; and hemochromatosis using serum iron, TIBC, ferritin and transferrin saturation. Each patient shall have an abdominal ultrasonography. UGI endoscopy would be done, if indicated.
5. Standard of Care Treatment:

   Standard of care treatment for patients with cirrhosis and overt acute encephalopathy shall be given to all patients.
   1. Identification of other potential causes for altered mental state i.e. head injury or drug intoxication shall be done.
   2. Identification and treatment of the precipitating causes of encephalopathy such as sepsis, gastrointestinal bleeding, hypokalemia (serum Potassium < 3.5mEq/L), alkalosis, azotemia, dehydration, diuretics, constipation, large protein intake and psychoactive drugs shall be done.
   3. Lactulose syrup: 30-120 ml in three divided doses through a nasogastric tube/ orally to produce 2-3 semi formed stools and/or lactulose retention enemas (300 ml lactulose +700 ml water) twice daily. No other ammonia lowering agent shall be given to these patients.
6. Monitoring and follow-up:

   Clinical Monitoring:

   All patients will be admitted to the intensive care unit/ high dependency unit, and shifted to ward once they revert back to grade I HE. Continuous monitoring of vital signs shall be done. Neurologic monitoring shall be done twice daily and grading of mental state will be as per the West Haven Criteria.

   Definition of Response to therapy:

   The assessment of the clinical response will be defined as follows:
   1. Resolution: disappearance of the HE clinical syndrome during the study
   2. Improvement: a decrease in the HE by 1 grade, but not reaching grade 0
   3. No Improvement: no improvement in HE
   4. Failure: shift to a higher grade of HE.

   Biochemical monitoring:

   Biochemical monitoring and monitoring of ammonia levels shall be done as mentioned above (under 'laboratory tests')

   Monitoring for Adverse Events:

   Any adverse event will be recorded specifying the time of onset, the duration, the severity and the relationship to the test medication.

   Tolerability: Tolerability of the study drug will be assessed by comparison of full blood cell count, liver function tests and renal function tests at baseline and at end of treatment.
7. End points:

   Primary end-point

   1. Completion of 5 days of treatment

   Secondary end-point
   1. Liver related death
   2. Death due to other causes
   3. Discontinuation due to adverse effects
   4. Discharge from hospital
8. Sample size: Sample size for this study was estimated using results of a previous study which reported complete recovery of encephalopathy in 79% patients in LOLA group and 55.6% patients in the placebo group (25). At 80% power and a 5% significance level (two-sided), 71 patients in each group would be required to detect a 22% difference in proportions. Assuming a dropout rate of 15% approximately (28), we will need to enroll 164 patients, i.e. 82 in each treatment arm.
9. Statistical Analysis: A chi-squared test will be used to compare the proportion of patients with complete reversal of HE after 5 days in LOLA treatment and placebo groups. A 95% confidence interval for the difference in proportions will also be calculated. A Chi-squared test will then be used to compare the HE grading at 5 days between the groups. Blood ammonia levels will be compared between groups using an independent samples t-test; while length of hospital stay is not expected to be normally distributed and therefore will be compared using a non-parametric Mann-Whitney test. All statistical tests will be 2-sided and using a 5% significance level.

ELIGIBILITY:
Inclusion Criteria:

* Hepatic cirrhosis based on clinical, biochemical, radiological and/or histological data
* Patients with overt acute grade 2, 3 and 4 HE, according to the West Haven criteria, with or without precipitating factors.
* Age of patient 18-70 years

Exclusion Criteria:

* Patients who are terminally ill
* Acute on chronic liver failure
* Hepatocellular carcinoma
* Wilson's disease as the etiological factor of liver disease
* Advanced cardiac or pulmonary disease
* Presence of underlying chronic renal failure
* Neuro-degenerative disease or major psychiatric illness
* Patients on sedatives or antidepressants
* Pregnancy or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Mental state grade | 5 days
  Mental state grade according to West Haven criteria for Hepatic encephalopathy

SECONDARY OUTCOMES:
Blood Ammonia levels | 5 days
  Change in blood ammonia levels will be measured at baseline and after 5 days of treatment
Mortality | 4 weeks
  Mortality rate in the two groups at 4 weeks will be compared
Length of Hospital stay | 4 weeks
  The total length of hospital stay (number of days) in each group will be compared.
Serum Cytokine levels | 5 days
  Change in serum cytokine levels (Interleukin-1, Interleukin-6, Interleukin-10 and TNF-alpha will be measured at baseline and after 5 days of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep S Sidhu, MD,DM, Principal Investigator — Professor, Dept of Gastroenterology, DMC and Hospital, Ludhiana, India; Omesh Goyal, MD, DM, Principal Investigator — Assistant Professor, Dept of Gastroenterology, DMC and Hospital, Ludhiana, India; B C Sharma, D.M., Principal Investigator — Professor, Dept of Gastroenterology, G.B. Pant Hospital, New Delhi
Locations (2):
- India (2):
  - G.B. Pant Hospital, New Delhi, New Delhi
  - Department of Gastroenterology, D.M.C. and Hospital, Ludhiana, Punjab

REFERENCES:
- [Background] Mas A. Hepatic encephalopathy: from pathophysiology to treatment. Digestion. 2006;73 Suppl 1:86-93. doi: 10.1159/000089783. Epub 2006 Feb 8. PMID 16498256
- [Background] Lizardi-Cervera J, Almeda P, Guevara L, Uribe M. Hepatic encephalopathy: a review. Ann Hepatol. 2003 Jul-Sep;2(3):122-30. PMID 15115963
- [Background] Groeneweg M, Moerland W, Quero JC, Hop WC, Krabbe PF, Schalm SW. Screening of subclinical hepatic encephalopathy. J Hepatol. 2000 May;32(5):748-53. doi: 10.1016/s0168-8278(00)80243-3. PMID 10845661
- [Background] Shawcross DL, Olde Damink SW, Butterworth RF, Jalan R. Ammonia and hepatic encephalopathy: the more things change, the more they remain the same. Metab Brain Dis. 2005 Sep;20(3):169-79. doi: 10.1007/s11011-005-7205-0. PMID 16167195
- [Background] Ferenci P, Lockwood A, Mullen K, Tarter R, Weissenborn K, Blei AT. Hepatic encephalopathy--definition, nomenclature, diagnosis, and quantification: final report of the working party at the 11th World Congresses of Gastroenterology, Vienna, 1998. Hepatology. 2002 Mar;35(3):716-21. doi: 10.1053/jhep.2002.31250. PMID 11870389
- [Background] Atluri DK, Prakash R, Mullen KD. Pathogenesis, diagnosis, and treatment of hepatic encephalopathy. J Clin Exp Hepatol. 2011 Sep;1(2):77-86. doi: 10.1016/S0973-6883(11)60126-6. Epub 2011 Nov 9. PMID 25755319
- [Background] Bajaj JS, Cordoba J, Mullen KD, Amodio P, Shawcross DL, Butterworth RF, Morgan MY; International Society for Hepatic Encephalopathy and Nitrogen Metabolism (ISHEN). Review article: the design of clinical trials in hepatic encephalopathy--an International Society for Hepatic Encephalopathy and Nitrogen Metabolism (ISHEN) consensus statement. Aliment Pharmacol Ther. 2011 Apr;33(7):739-47. doi: 10.1111/j.1365-2036.2011.04590.x. Epub 2011 Feb 9. PMID 21306407
- [Background] Shawcross D, Jalan R. Dispelling myths in the treatment of hepatic encephalopathy. Lancet. 2005 Jan 29-Feb 4;365(9457):431-3. doi: 10.1016/S0140-6736(05)17832-5. PMID 15680459
- [Background] Ferenci P, Herneth A, Steindl P. Newer approaches to therapy of hepatic encephalopathy. Semin Liver Dis. 1996 Aug;16(3):329-38. doi: 10.1055/s-2007-1007245. No abstract available. PMID 8989818
- [Background] Uribe M, Moran S, Poo JL, Mendez-Sanchez N, Guevara L, Garcia-Ramos G. Beneficial effect of carbohydrate maldigestion induced by a disaccharidase inhibitor (AO-128) in the treatment of chronic portal-systemic encephalopathy. A double-blind, randomized, controlled trial. Scand J Gastroenterol. 1998 Oct;33(10):1099-106. doi: 10.1080/003655298750026822. PMID 9829367
- [Background] Als-Nielsen B, Gluud LL, Gluud C. Non-absorbable disaccharides for hepatic encephalopathy: systematic review of randomised trials. BMJ. 2004 May 1;328(7447):1046. doi: 10.1136/bmj.38048.506134.EE. Epub 2004 Mar 30. PMID 15054035
- [Background] Bongaerts G, Severijnen R, Timmerman H. Effect of antibiotics, prebiotics and probiotics in treatment for hepatic encephalopathy. Med Hypotheses. 2005;64(1):64-8. doi: 10.1016/j.mehy.2004.07.029. PMID 15533613
- [Background] Paik YH, Lee KS, Han KH, Song KH, Kim MH, Moon BS, Ahn SH, Lee SJ, Park HJ, Lee DK, Chon CY, Lee SI, Moon YM. Comparison of rifaximin and lactulose for the treatment of hepatic encephalopathy: a prospective randomized study. Yonsei Med J. 2005 Jun 30;46(3):399-407. doi: 10.3349/ymj.2005.46.3.399. PMID 15988813
- [Background] Mas A, Rodes J, Sunyer L, Rodrigo L, Planas R, Vargas V, Castells L, Rodriguez-Martinez D, Fernandez-Rodriguez C, Coll I, Pardo A; Spanish Association for the Study of the Liver Hepatic Encephalopathy Cooperative Group. Comparison of rifaximin and lactitol in the treatment of acute hepatic encephalopathy: results of a randomized, double-blind, double-dummy, controlled clinical trial. J Hepatol. 2003 Jan;38(1):51-8. doi: 10.1016/s0168-8278(02)00350-1. PMID 12480560
- [Background] Riordan SM, Williams R. Treatment of hepatic encephalopathy. N Engl J Med. 1997 Aug 14;337(7):473-9. doi: 10.1056/NEJM199708143370707. No abstract available. PMID 9250851
- [Background] Rose C, Michalak A, Pannunzio P, Therrien G, Quack G, Kircheis G, Butterworth RF. L-ornithine-L-aspartate in experimental portal-systemic encephalopathy: therapeutic efficacy and mechanism of action. Metab Brain Dis. 1998 Jun;13(2):147-57. doi: 10.1023/a:1020613314572. PMID 9699922
- [Background] Staedt U, Leweling H, Gladisch R, Kortsik C, Hagmuller E, Holm E. Effects of ornithine aspartate on plasma ammonia and plasma amino acids in patients with cirrhosis. A double-blind, randomized study using a four-fold crossover design. J Hepatol. 1993 Nov;19(3):424-30. doi: 10.1016/s0168-8278(05)80553-7. PMID 8151104
- [Background] Kircheis G, Nilius R, Held C, Berndt H, Buchner M, Gortelmeyer R, Hendricks R, Kruger B, Kuklinski B, Meister H, Otto HJ, Rink C, Rosch W, Stauch S. Therapeutic efficacy of L-ornithine-L-aspartate infusions in patients with cirrhosis and hepatic encephalopathy: results of a placebo-controlled, double-blind study. Hepatology. 1997 Jun;25(6):1351-60. doi: 10.1002/hep.510250609. PMID 9185752
- [Background] Stauch S, Kircheis G, Adler G, Beckh K, Ditschuneit H, Gortelmeyer R, Hendricks R, Heuser A, Karoff C, Malfertheiner P, Mayer D, Rosch W, Steffens J. Oral L-ornithine-L-aspartate therapy of chronic hepatic encephalopathy: results of a placebo-controlled double-blind study. J Hepatol. 1998 May;28(5):856-64. doi: 10.1016/s0168-8278(98)80237-7. PMID 9625322
- [Background] Rees CJ, Oppong K, Al Mardini H, Hudson M, Record CO. Effect of L-ornithine-L-aspartate on patients with and without TIPS undergoing glutamine challenge: a double blind, placebo controlled trial. Gut. 2000 Oct;47(4):571-4. doi: 10.1136/gut.47.4.571. PMID 10986219
- [Background] Chen MF, Li RC, Chen CH, Gao XC. [Therapeutic effect of L-ornithine-L-aspartate on liver cirrhosis complicated by hepatic encephalopathy]. Di Yi Jun Yi Da Xue Xue Bao. 2005 Jun;25(6):718-9, 722. Chinese. PMID 15958319
- [Background] Poo JL, Gongora J, Sanchez-Avila F, Aguilar-Castillo S, Garcia-Ramos G, Fernandez-Zertuche M, Rodriguez-Fragoso L, Uribe M. Efficacy of oral L-ornithine-L-aspartate in cirrhotic patients with hyperammonemic hepatic encephalopathy. Results of a randomized, lactulose-controlled study. Ann Hepatol. 2006 Oct-Dec;5(4):281-8. PMID 17151582
- [Background] Abdo-Francis JM, Perez-Hernandez JL, Hinojosa-Ruiz A, Hernandez-Vasquez JR. [Reduction of hospital stay with the use of L-ornithine L-aspartate (LOLA) in patients with hepatic encephalopathy]. Rev Gastroenterol Mex. 2010;75(2):135-41. Spanish. PMID 20615780
- [Background] Ahmad I, Khan AA, Alam A, Dilshad A, Butt AK, Shafqat F, Malik K, Sarwar S. L-ornithine-L-aspartate infusion efficacy in hepatic encephalopathy. J Coll Physicians Surg Pak. 2008 Nov;18(11):684-7. PMID 18983791
- [Background] Kircheis G, Wettstein M, Dahl Sv, Haussinger D. Clinical efficacy of L-ornithine-L-aspartate in the management of hepatic encephalopathy. Metab Brain Dis. 2002 Dec;17(4):453-62. doi: 10.1023/a:1021934607762. PMID 12602521
- [Background] Jiang Q, Jiang XH, Zheng MH, Chen YP. L-Ornithine-l-aspartate in the management of hepatic encephalopathy: a meta-analysis. J Gastroenterol Hepatol. 2009 Jan;24(1):9-14. doi: 10.1111/j.1440-1746.2008.05582.x. Epub 2008 Sep 24. PMID 18823442
- [Background] Acharya SK, Bhatia V, Sreenivas V, Khanal S, Panda SK. Efficacy of L-ornithine L-aspartate in acute liver failure: a double-blind, randomized, placebo-controlled study. Gastroenterology. 2009 Jun;136(7):2159-68. doi: 10.1053/j.gastro.2009.02.050. PMID 19505424
- [Background] Goggs R, Serrano S, Szladovits B, Keir I, Ong R, Hughes D. Clinical investigation of a point-of-care blood ammonia analyzer. Vet Clin Pathol. 2008 Jun;37(2):198-206. doi: 10.1111/j.1939-165X.2008.00024.x. PMID 18533920